CLINICAL TRIAL: NCT01145638
Title: A Phase III, Randomized, Open-label Study of Intravenous Iron Isomaltoside 1000 (Monofer®) as Mono Therapy (Without Erythropoiesis Stimulating Agents) in Comparison With Oral Iron Sulfate in Subjects With Non-myeloid Malignancies Associated With Chemotherapy Induced Anaemia (CIA)
Brief Title: A Study of Intravenous Iron Isomaltoside 1000 (Monofer®) as Mono Therapy (Without Erythropoiesis Stimulating Agents) in Comparison With Oral Iron Sulfate in Subjects With Non-myeloid Malignancies Associated With Chemotherapy Induced Anaemia (CIA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P-Monofer-CIA-01; EudraCT no. 2009-016727-53
Record Dates: First submitted 2010-06-15; First posted 2010-06-16 (Estimated); Results first posted 2015-12-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-04

CONDITIONS: Non-myeloid Malignancies; Chemotherapy Induced Anaemia
Keywords: cancer; chemotherapy induced anaemia; iron; Patients with non-myeloid malignancies and Chemotherapy Induced Anaemia (CIA); CIA
MeSH Terms: conditions — Neoplasms | interventions — iron isomaltoside 1000; Iron-Dextran Complex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- iron isomaltoside 1000 (Experimental): Iron isomaltoside intravenously as bolus or infusion
  Interventions: Drug: iron isomaltoside 1000
- iron sulphate (Active Comparator): oral iron sulphate twice a day
  Interventions: Drug: iron sulphate

INTERVENTIONS:
Drug: iron isomaltoside 1000 — intravenously as bolus or infusion, 500 mg or 1000mg up to full replacement dose
  Other Names: Monofer
  Arms: iron isomaltoside 1000
Drug: iron sulphate — oral, 200 mg per day (100 mg bid),12 weeks
  Other Names: Ferroduretter
  Arms: iron sulphate

SUMMARY:
The purpose of this study is to compare the efficacy and safety of intravenous iron therapy with oral iron therapy in patients with cancer and chemotherapy induced anaemia.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged more than 18 years.
2. Subjects diagnosed with cancer (non-myeloid malignancies) receiving chemotherapy at least 1 day prior to screening and who are going to receive at least two more chemotherapy cycles.
3. Hb < 12 g/dL (7.4 mmol/L).
4. TfS <50%.
5. Serum Ferritin <800 ng/ml.
6. An Eastern Cooperative Oncology Group (ECOG) performance status of 0 to
7. Willingness to participate after informed consent (including HIPAA, if applicable).

Exclusion Criteria:

1. Anemia caused primarily by other factors than CIA.
2. IV or oral iron treatment within 4 weeks prior to screening visit.
3. Erythropoietin treatment within 4 weeks prior to screening visit.
4. Blood transfusion within 4 weeks prior to screening visit.
5. Imminent expectation of blood transfusion on part of treating physician.
6. Iron overload or disturbances in utilization of iron (e.g. haemochromatosis and haemosiderosis).
7. Drug hypersensitivity (i.e. previous hypersensitivity to Iron Dextran or iron mono- or disaccharide complexes or to iron sulfate).
8. Known hypersensitivity to any excipients in the investigational drug products.
9. Subjects with a history of multiple allergies.
10. Decompensated liver cirrhosis or active hepatitis (alanine aminotransferase (ALAT) > 3 times upper normal limit).
11. Active acute or chronic infections (assessed by clinical judgement and if deemed necessary by investigator supplied with white blood cells (WBC) and C-reactive protein (CRP)).
12. Rheumatoid arthritis with symptoms or signs of active joint inflammation.
13. Pregnancy and nursing (To avoid pregnancy, women have to be postmenopausal (at least 12 months must have elapsed since last menstruation), surgically sterile, or women of child bearing potential must use one of the following contraceptives during the whole study period and after the study has ended for at least 5 times plasma biological half-life of the investigational medicinal product: Contraceptive pills, intrauterine devices (IUD), contraceptive depot injections (prolonged-release gestagen), subdermal implantation, vaginal ring, and transdermal patches).
14. Planned elective surgery during the study.
15. Participation in any other clinical study (except chemotherapy protocol) within 3 months prior to screening.
16. Known intolerance to oral iron treatment.
17. Untreated B12 or folate deficiency.
18. Any other medical condition that, in the opinion of Principal Investigator, may cause the subject to be unsuitable for the completion of the study or place the subject at potential risk from being in the study. Example, Uncontrolled Hypertension, Unstable Ischemic Heart Disease or Uncontrolled Diabetes Mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2010-10; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Lykke Thomsen, MD, Study Chair — Pharmacosmos A/S
Locations (1):
- Apollo Hospitals, New Delhi, India

REFERENCES:
- [Derived] Birgegard G, Henry D, Glaspy J, Chopra R, Thomsen LL, Auerbach M. A Randomized Noninferiority Trial of Intravenous Iron Isomaltoside versus Oral Iron Sulfate in Patients with Nonmyeloid Malignancies and Anemia Receiving Chemotherapy: The PROFOUND Trial. Pharmacotherapy. 2016 Apr;36(4):402-14. doi: 10.1002/phar.1729. Epub 2016 Apr 1. PMID 26927900

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Iron Isomaltoside 1000 | Iron Sulphate
Started | 231 | 119
Completed | 141 | 62
Not Completed | 90 | 57

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Iron Isomaltoside 1000 | Iron Sulphate | Total
Number analyzed (Participants) | 231 | 119 | 350
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 187 | 101 | 288
  >=65 years | 44 | 18 | 62
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 90 | 241
  Male | 80 | 29 | 109
Region of Enrollment [Number; unit: participants]
  India | 133 | 72 | 205
  Germany | 7 | 3 | 10
  Denmark | 3 | 1 | 4
  Spain | 2 | 0 | 2
  Poland | 40 | 16 | 56
  Russian Federation | 29 | 18 | 47
  Sweden | 5 | 3 | 8
  United States | 12 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Hb Concentration
Time Frame: Baseline week 4
Population: The FAS population included all the subjects who were randomised into the study, received at least one dose of the study drug, and had at least one post-baseline Hb assessment. The subjects were considered as randomised, regardless of which treatment they actually received.
Measure: Mean (Full Range); unit: g/dL
Arm/Group | Iron Isomaltoside 1000 | Iron Sulphate
Number analyzed (Participants) | 192 | 99
g/dL | 0.48 [-4 to 4] | 0.44 [-2 to 4]

2. Secondary Outcome: Change in Hemoglobin From Baseline to Week 24
Time Frame: 24 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: g/dL
Arm/Group | Iron Isomaltoside 1000 | Iron Sulphate
Number analyzed (Participants) | 157 | 72
g/dL | 1.60 [-6.3 to 6.5] | 1.78 [-5.3 to 7.4]

ADVERSE EVENTS:
Description: The safety population included all subjects who were randomised and received at least one dose of iron isomaltoside 1000 or iron sulphate. The safety analyses was performed on the safety population.
Arm/Group | Iron Isomaltoside 1000 | Iron Sulphate
Serious Adverse Events (participants affected / at risk) | 32/229 | 18/112
Other Adverse Events (participants affected / at risk) | 173/229 | 107/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iron Isomaltoside 1000 (N=229) | Iron Sulphate (N=112)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1)
Sudden death (General disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Unirary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (9) | 7 (7)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoe (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iron Isomaltoside 1000 (N=229) | Iron Sulphate (N=112)
Anaemia (Blood and lymphatic system disorders) | 20 (22) | 12 (13)
Leukopenia (Blood and lymphatic system disorders) | 12 (13) | 10 (13)
Neutropenia (Blood and lymphatic system disorders) | 15 (21) | 6 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (13) | 7 (11)
Constipation (Gastrointestinal disorders) | 7 (8) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 8 (14) | 10 (11)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 9 (9)
Nausea (Gastrointestinal disorders) | 14 (19) | 8 (12)
Stomatitis (Gastrointestinal disorders) | 14 (14) | 5 (5)
Vomiting (Gastrointestinal disorders) | 16 (24) | 7 (8)
Asthenia (General disorders) | 18 (20) | 7 (9)
Pyrexia (General disorders) | 12 (13) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 17 (17) | 9 (9)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If Pharmacosmos or its agents has not prepared a draft for submission to a peer reviewed journal prior to 1 year following completion of the study report, the investigators have the right to publish the results. Such publications are to be submitted to Pharmacosmos for comment 30 days prior to submission for publication.